CLINICAL TRIAL: NCT02420886
Title: The Effects of GM-CSF, HB-EGF and LIF Cytokines Supplementation Need Verification for Human Embryo Development in Vitro
Brief Title: Adding Cytokines to In Vitro Human Culture Media to Improve Embryogenesis and Implantation
Acronym: GHLCSHED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banon IVF Center Assiut, Egypt (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Laboratory Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Ibnsina IVF center
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Infertility
Keywords: In Vitro culture of human embryos
MeSH Terms: conditions — Infertility | interventions — Heparin-binding EGF-like Growth Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cytokines supplemented In Vitro single culture media (Active Comparator): We will add Cytokines (LIF, HB-EGF and GM-CSF) to LIFEGLOBAL culture media and assess the embryogenesis and pregnancy.
  Interventions: Other: Adding LIF, HB-EGF and GM-CSF to Lifeglobal human IVF culture media
- Traditional Single step culture media (No Intervention)

INTERVENTIONS:
Other: Adding LIF, HB-EGF and GM-CSF to Lifeglobal human IVF culture media
  Arms: Cytokines supplemented In Vitro single culture media

SUMMARY:
Assessment of the embryological benefit of in vitro adding of Cytokines (LIF 5ng/ml, HB-EGF 5ng/ml and GM-CSF 2n/ml) to the culture media and closely monitor its effect on embryogenesis and implantation outcomes.

DETAILED DESCRIPTION:
The IVF culture media design and upgrade underwent many ideas during the last 3 decades, we suppose that adding the Cytokines (LIF 5ng/ml, HB-EGF 5ng/ml and GM-CSF 2ng/ml) as a growth factor that have multi-ways to might improve embryo development in vitro so we decide to design a trial to compare the embryogenesis by sibling Oocytes of the same patient between two arm of the same culture media and the same culture condition. One arm with Cytokines and the other is traditional one and closely monitor the outcome within the 2 arms and record the results.

ELIGIBILITY:
Inclusion Criteria:

* all patients

Exclusion Criteria:

* over 40 years

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 443 (Actual)
Dates: Start 2015-05-16 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate ( % ) | 6 months

SECONDARY OUTCOMES:
clinical pregnancy rate ( % ) | 6 months
implantation rate | 6 months
fertilization rate | 6 days of culture
top-quality embryo rate | 6 days of culture
rates for blastocyst formation and quality | 6 days of culture
embryo utilization rate | 6 days of culture

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Banon IVF Center, Asyut
  - Ibnsina IVF center, Sohag

REFERENCES:
- [Derived] Fawzy M, Emad M, Elsuity MA, Mahran A, Abdelrahman MY, Fetih AN, Abdelghafar H, Sabry M, Nour M, Rasheed SM. Cytokines hold promise for human embryo culture in vitro: results of a randomized clinical trial. Fertil Steril. 2019 Nov;112(5):849-857.e1. doi: 10.1016/j.fertnstert.2019.07.012. Epub 2019 Sep 21. PMID 31551154